CLINICAL TRIAL: NCT04611841
Title: Medical-biological Research of the Pathogenesis of Disease Caused by SARS-CoV-2
Brief Title: Medical-biological Research of the Pathogenesis of COVID-19 Disease Caused by SARS-CoV-2
Acronym: COV2020
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Federal Research and Clinical Center of Physical-Chemical Medicine (Other)
Collaborators: Burnasyan Federal Medical Biophysical Center (Other Government); Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government); Moscow city hospital named after S.I. Spasokukotskiy (Unknown); Federal State Public Scientific Institution, Scientific Center for Family Health and Human Reproduction Problems (Other); Federal State Budgetary Healthcare Institution, Hospital RAS (Unknown)
Responsible Party: Sponsor
Other Study IDs: COV2020
Record Dates: First submitted 2020-09-26; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Covid19
Keywords: Metavirome; SARS-CoV-2; Pathogenesis; Oxidative stress; Peptides
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Сonducting in-depth medical and biological studies of the pathogenesis of the disease caused by the SARS-CoV-2 in Moscow, the Moscow region and some other regions of the Russian Federation.

DETAILED DESCRIPTION:
To date, none of the methods used to test for coronavirus infection provide reliable information about the status of an individual's infection. Common tests based on PCR, carried out on the basis of samples taken from the human respiratory tract, give a positive answer in far from all cases. Antibody tests may not record the initial stages of the disease, or may not reveal residual immunity in those who have been ill, while giving cross-reactions to other common coronaviruses.

A comprehensive assessment of the biological parameters of the virus and the parameters of the immune response to infection is required. In this regard, we propose an integrated approach, including the use of PCR testing technology, analysis of the immune response in the form of antibodies of all major classes (IgG, IgA), determination of inflammation markers, C-reactive protein, detailed blood test, ferritin and troponin.

In addition, an analysis of the genetic diversity of strains of the pathogen COVID-19 circulating among various groups of the population of the Russian Federation will be carried out.

To collect and analyze data, it is planned to enter information into a special electronic system and analyze the collected data with a wide range of informative methods that allow "layer by layer" to compare and collect a complete picture of what is happening.

Objectives of the study:

1. Identifying the percentage of infected in the population in Moscow, the Moscow region and some other regions where the epidemic situation in connection with SARS-CoV-2 remains tense;
2. Study of genetic diversity (including metavirome) and dynamics of structural variability of the causative agent of coronavirus infection in the studied regions;
3. Studying the features of the formation and tension of immunity in patients who have undergone coronavirus infection of varying severity;
4. Clarification of the mechanisms of occurrence and development of coronavirus infection.

In the study of biological samples obtained from research participants, methods of proteomics, peptidomics, next generation sequencing (NGS), physicochemical methods of analysis will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 and under 75 years old
* COVID-19 diagnosis confirmed by PCR test
* Written consent to participate in the study

Exclusion Criteria:

* Unwillingness or inability to give written informed consent to participate in the study
* A serious condition with a threat to life or contraindications that prevent the collection of biomaterial
* Oncological diseases outside the stage of remission

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mostly urban residents, at least 18 years old and no more than 75 years old with clinical manifestations and laboratory confirmed new coronavirus infection.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Determination of antibody binding of patients diagnosed with COVID-19 to proteins of the SARS-CoV-2 virus | Through samples collection end, an average of 2 years
  Visualization of antibody binding to linear and volumetric sequences SARS-CoV-2 proteins of the virus in 200 samples of blood plasma by the methods Western blot and enzyme-linked immunosorbent assay. It is necessary to identify the epitopes of the SARS-CoV-2 virus recognized by the human immune system and to analyze the individual response of different patients to coronavirus infection.
  Sample collection time points: Point 1 - on the day of admission if there is a positive test for RNA virus or on the day of receipt of confirmation of the presence of the virus in an already hospitalized patient; Point 6 - an acute condition, regardless of the day of observation; Point 7 - statement, regardless of the day of observation.
Determination of the presence of peptides of the SARS-CoV-2 virus in the plasma of patients diagnosed with COVID-19 | Through samples collection end, an average of 2 years
  Determination of the presence of peptides of the SARS-CoV-2 virus in 100 samples of blood plasma, confirmed by mass spectrometry. It is necessary to identify the correlation between the severity of the coronavirus infection and the presence of viral peptides in the patient's blood
  Sample collection time points: Point 1 - on the day of admission if there is a positive test for RNA virus or on the day of receipt of confirmation of the presence of the virus in an already hospitalized patient; Point 6 - an acute condition, regardless of the day of observation; Point 7 - statement, regardless of the day of observation.
Determination of the degree of oxidative damage to lipids (lipid peroxidation) in the blood plasma of patients infected with coronavirus | Through samples collection end, an average of 2 years
  The content of lipid peroxidation products in blood plasma, expressed in μg / ml of plasma.
  Analysis 200 samples of blood plasma by spectrophotometric and spectrofluorimetric methods. To demonstrate a statistically significant difference from the control group of patients not infected with coronavirus.
  Sample collection time points: Point 1 - on the day of admission if there is a positive test for RNA virus or on the day of receipt of confirmation of the presence of the virus in an already hospitalized patient; Point 6 - an acute condition, regardless of the day of observation; Point 7 - statement, regardless of the day of observation.
Revealing the degree of protein damage in the blood plasma of patients infected with coronavirus | Through samples collection end, an average of 2 years
  The content of average weight molecules in blood plasma, expressed in μg / ml of plasma.
  Analysis 200 samples of blood plasma by spectrophotometric method. To demonstrate a statistically significant difference from the control group of patients not infected with coronavirus.
  Sample collection time points: Point 1 - on the day of admission if there is a positive test for RNA virus or on the day of receipt of confirmation of the presence of the virus in an already hospitalized patient; Point 6 - an acute condition, regardless of the day of observation; Point 7 - statement, regardless of the day of observation.
Measurement of iron (Fe3+) content in blood plasma of patients infected with coronavirus | Through samples collection end, an average of 2 years
  The content of iron ions (Fe3+) in units of optical density per 1 ml of plasma. Analysis 200 samples of blood plasma by spectrophotometric method. To demonstrate a statistically significant difference from the control group of patients not infected with coronavirus.
  Sample collection time points: Point 1 - on the day of admission if there is a positive test for RNA virus or on the day of receipt of confirmation of the presence of the virus in an already hospitalized patient; Point 6 - an acute condition, regardless of the day of observation; Point 7 - statement, regardless of the day of observation.
Metagenomic analysis of viral and bacterial respiratory flora of selected samples | Through samples collection end, an average of 2 years
  500 metagenomes for comparative bioinformatics analysis of viral and bacterial flora in patients with COVID-19 of varying severity.
  Sample collection time points: Point 1 - on the day of admission if there is a positive test for RNA virus or on the day of receipt of confirmation of the presence of the virus in an already hospitalized patient; Point 6 - an acute condition, regardless of the day of observation; Point 7 - statement, regardless of the day of observation.
Analysis of the genetic variability of the SARS-CoV-2 virus, including the heterogeneity of the viral population in one patient | Through samples collection end, an average of 2 years
  Bioinformatic analysis of the 500 viral genomes for comparison genetic characteristics of different strains SARS-CoV-2.
  Sample collection time points: Point 1 - on the day of admission if there is a positive test for RNA virus or on the day of receipt of confirmation of the presence of the virus in an already hospitalized patient; Point 6 - an acute condition, regardless of the day of observation; Point 7 - statement, regardless of the day of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Vadim Govorun, MD, Study Director — FRCC PCM
Locations (1):
- Federal Research and Clinical Center of Physical-Chemical Medicine of Federal Medical Biological Agency, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided